CLINICAL TRIAL: NCT07030387
Title: Evaluation of the Effectiveness of a Very Brief Smoking Cessation Intervention in Family Health Centers: A Pragmatic Randomized Controlled Trial
Brief Title: Evaluation of the Effectiveness of a Very Brief Smoking Cessation Intervention in Family Health Centers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Yigit Yagci, Family Medicine Specialist, MD, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/217
Record Dates: First submitted 2025-06-05; First posted 2025-06-22 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Smoking Cessation; Tobacco Dependence
Keywords: Smoking cessation; Primary health care; Pragmatic clinic trials; Randomized controlled trial; Motivation; Health behavior
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder; Health Behavior

STUDY DESIGN:
Intervention Model Description: 3A-OR Model (Ask - Assess - Advise - Offer Assistance - Record) In this brief intervention algorithm, the physician primarily learns every patient's smoking status, assesses the smoker's motivation to quit, advises cessation with different approaches for the pre-contemplation and contemplation/preparation stages, then offers assistance, and finally records the encounter in the patient's file.
  1. (A) LEARN!
  2. (A) ASSESS!
     If the smoker is in the PRE-CONTEMPLATION stage:
  3. (A) ADVISE!
  4. (O) OFFER ASSISTANCE!
  5. (R) RECORD!
  If the smoker is in the CONTEMPLATION or PREPARATION stage:
  3. (A) ADVISE! 4. (O) OFFER ASSISTANCE! 5. (R) RECORD!
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3A-OR very brief smoking cessation intervention (Experimental): Patients of family physicians who had begun implementing 3A-OR very brief smoking cessation intervention as their routine clinical practices constituted the intervention group of the trial.
  Interventions: Behavioral: Smoking cessation counselling group
- Control group: same-day patients of other family physicians in the same Family Health Centers (Experimental): Patients of the other family physicians in the same family health centers were assigned to the control group.
  Interventions: Behavioral: Control group patients were those who had not received the 3A-OR intervention

INTERVENTIONS:
Behavioral: Smoking cessation counselling group — 3A-OR very brief intervention for smoking cessation
  Arms: 3A-OR very brief smoking cessation intervention
Behavioral: Control group patients were those who had not received the 3A-OR intervention — Control Group (Patients of the other family physicians in the same family health centers)
  Arms: Control group: same-day patients of other family physicians in the same Family Health Centers

SUMMARY:
In Turkey, the prevalence of tobacco use among individuals was 31.4% in 2019. The WHO recommends brief and very brief interventions to increase tobacco cessation rates and medical support. In developing countries, these brief interventions are being integrated into primary care. The aim of this study is to evaluate the effectiveness of very brief interventions at different family health centers in Aydın province.

A pragmatic randomized controlled trial was conducted with 170 patients in intervention group and 161 in control group across 14 family health centers in Aydın province from June 2023 to December 2023. Physicians that recurited for intervention received one hour of online training before applying very brief smoking cessation interventions to their patients. Data collection included a baseline assessment of sociodemographic characteristics, smoking status, and medical history. At the three-month follow-up, participants' cessation status and motivations were assessed via phone call interviews. Intention to Treat approach was utilized. Secondary outcomes included the objective and subjective frequency of smoking, as well as treatment and support received.

DETAILED DESCRIPTION:
INTRODUCTION:

Tobacco use is among the leading causes of preventable mortality. One in ten deaths is related to tobacco use worldwide. Expected lifespan of smokers is ten years shorter than non-smokers and half of them lose around 20 Quality-Adjusted Life Years (QALYs) due to tobacco related diseases before death.

The motto "Offer help to quit tobacco use" has the worst progression within MPOWER strategies of WHO. Smoking cessation services are especially inadequate in developing countries, and even when offered free of charge, their utilisation rates remain low.

On the other hand, brief physician advice enhances the quitting rates of smokers. WHO recommends brief clinical interventions to enhance tobacco cessation rates. Former studies show that these interventions increase the cessation rates. A meta-analysis specifically examining brief interventions integrated into primary care setting has found that they effectively improve smoking cessation rates. Therefore, authors suggest that behavioural healthcare services should be integrated into primary care to promote tobacco cessation intervention.

However, these interventions, which WHO defines as "brief", last 3-10 minutes and are difficult to implement in busy clinical practice settings where the time is allocated to a patient is limited. Lack of time and poor education are the main barriers to physicians using these interventions efficiently.

To increase physicians' adherence, very brief interventions (30-60 seconds) are also recommended. AAR (Ask-Advice-Refer) brief intervention, which has been developed based on 5A approach, prioritises increasing awareness, advice and referral. AAC (Ask-Advice-Connect) approach which aims to increase the uptake of referral smokers to smoking cessation counseling services is also recommended. AWARD (Ask-Warn-Advice-Refer-Do it again) and WAR (Warn-Advice-Refer) models emphasise the warning that "one in every two smokers dies because of smoking". These very brief interventions do not focus on smokers' motivation to quit. The 3A-OR very brief intervention which is conducted in family health centers consists of the steps "Ask-Assess-Advice-Offer-Record". This intervention primarily evaluates smokers' motivation of quit and can be tailored according to smoker's motivation level.

Studies evaluating the effectiveness and feasibility of very brief interventions are limited, with outcomes from only three recent studies to date. Nevertheless, these studies are mostly explanatory RCT's and have been conducted in hospitals.

In Türkiye, RCTs on this topic appear highly limited. The trial of the effectiveness of an intervention emphasising "Harm effects of Second hand tobbacco exposure on their children" to smoker mothers has been conducted in tertiary care hospital in 2006. Implementation and effectiveness of very brief smoking cessation interventions in primary care settings are unknown.

This study aims to evaluate effectiveness of 3A-OR very brief smoking cessation intervention in improving motivation levels and increasing quit rates of smokers in routine primary care practices.

METHODS:

Study design:

This paralelled multi-site pragmatic randomized controlled trial recruited smokers from 17 family health centers in primary care in the city of Aydın, Türkiye, from June 2023 to December 2023.

Ethical approval was granted by Ethics Committee of Adnan Menderes University Medical School. Written informed consent was obtained from participants who agreed to take part in the study after declaration the aim of study. Their contact information was kept confidential.

Recruitment procedures:

Family physicians working in primary care in the city of Aydın were invited for participating in a trial. Twenty voluntary family physicians from 17 family health centers were included in the intervention arm of the trial.

All (smoking) patients who attended 17 family health centers from June 2023 to December 2023 were eligible for the trial.

Randomization (Participants):

The study was carried out in two phases. In the first phase, physicians who accepted to take part in the intervention group received one-hour online training on the intervention, in May 2023. Participant physicians were informed by study team about 3A-OR very brief smoking cessation advice that can be applied in 30-60 seconds. Additionally, a few documents that contain detailed information on intervention and brochures for distribution to smoking patients were shared with the physicians. Regardless of their previous practices, physicians were required to develop an approach to evaluating their patients' smoking habits in accordance with 3A-OR intervention. It was highlighted that 3A-OR very brief smoking cessation intervention was expected become a part of their daily routine clinical practices.

In second phase, data were collected between June-December 2023. In this period, a member of research team (YY) visited Family Health Centers of the physicians in the intervention arm, according to a pre-determined schedule. He invited smoking patients to participate in the study just after completing the consultation with their family physicians in waiting rooms of the health centers. Within the framework of the study protocol, patients of family physicians who had begun implementing 3A-OR very brief smoking cessation intervention as their routine clinical practices constituted the intervention group of the trial. Patients of the other family physicians in the same family health centers were assigned to the control group.

Before the study, power analysis was performed using one-way Fisher's Exact test in the Gpower software. In three-month follow up, with an anticipated abstinance rate of 15% in last 7 days in the intervention group (%5 in the control group) to create an effect size of %10, the sample size was calculated as 126 from each group and 252 in total. Based on the estimated number of smoking patients per single working day, it was aimed to include at least 10 smokers for each of 20 family physicians in the intervention group, targeting 200 smokers per group and 400 smokers in total. Eligible smokers were consecutively recruited without using any systematic or randomised sampling.

Intervention:

Physicians in the intervention arm applied the intervention of 3A-OR protocol that was developed by the research team. That protocol includes the stages of "Ask-Assess-Advice-Offer-Record". Further details of this intervention are provided in the Appendix.

The investigators assumed that physicians in the intervention group delivered very brief intervention about smoking cessation to all of their patients, but physicians in control group did not deliver such an intervention. Nevertheless, physicians in control group might have talked about smoking cessation with their patients as a part of their usual patient-physician relations.

Baseline and follow-up data collection:

Baseline data were collected by the same researcher in the waiting rooms of family health centers where the study was conducted. There was no follow-up contact during study period of three month for additional data collection. However, if participants revisited their doctors, that physician could repeat the intervention. Three months after first face-to-face interview, the follow-up data were collected via phone calls by the same researcher.

Participants who completed interview with their physicians of either group filled out data collection form together with the researcher, without knowing which group they appointed to. Participants were informed about study at minimal level with considering ethical concerns, so as unaware about current intervention. Participants who did not aware of their group situation were assigned according to the group of their family physician. Thus, participants were randomized to intervention or control group in accordance with their family physicians at baseline contact. In this respect, study was conducted in a single-blind design.

Study data were collected via questionnaire form which was developed for the purpose. The questionnaire consisted of 8 questions covering sociodemographic characteristics at first contact, 10 questions assessing smoking related characteristics and 11 questions determining their general health status. The level of nicotine addiction was determined using the short version of Fagerstrom Test for Nicotine Dependence (FTND).

Outcomes:

The trial had two main outcomes. Primarily, successful quitting defined as participants' abstinence from smoking for at least a week at the end of three months. Observed motivation change to quit of participant smokers was the secondary outcome.

Sociodemographic, medical and baseline smoking-related characteristics in the questionnaire were the independent variables of the trial.

Statistical analysis:

Statistical analyses were performed using SPSS 22.0 statistical software package. Descriptive analysis included percentages, means and standard deviations; the normality of data distribution was assessed with Kolmogorov-Smirnov test. For comparative assessment between groups, Pearson Chi-Square test, Fisher's Exact test, Cochran-Mantel-Haenszel test, Log-Linear test were conducted for categorical variables and Mann-Whitney U test, Kruskal-Wallis test, Wilcoxon test were applied for continuous variables. Binary Logistic Regression was performed to determine possible confounders. P values <0.05 was considered statistically significant.

Study design was guided by the PRECIS-2 (Pragmatic-Explanatory Continuum Indicator Summary) tool framework.

ELIGIBILITY:
Inclusion Criteria:

* All smokers aged 18 and above who visited selected Family Health Centers

Exclusion Criteria:

* Smokers experiencing cooperation and communication issues
* Smokers who have received support for a smoking cessation attempt within the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Smoking Quit Rates | 3 months after the 3A-OR very brief intervention
  Smoking cessation rates between groups at 3 months follow up

SECONDARY OUTCOMES:
Motivational stages of quitting smoking | 3 months after the 3A-OR very brief intervention
  Smokers' motivational stage of quit smoking assessment with Prochaska's Transtheoretical Model (Stages of Change: Pre-contemplation, Contemplation, Preparation, Action, and Maintenance) in both the intervention and control groups at baseline and at the 3-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Okay BAŞAK, MD, PhD, Study Chair — Aydın Adnan Menderes University, School of Medicine, Department of Family Medicine; Melda DİBEK, MD, PhD, Study Director — Aydın Adnan Menderes University, School of Medicine, Department of Family Medicine; Yiğit YAĞCI, MD, Principal Investigator — Aydın Adnan Menderes University, School of Medicine, Department of Family Medicine
Locations (1):
- Assigned Family Health Centers within Aydin Province, Efeler, Aydın, Turkey (Türkiye)

REFERENCES:
- [Background] Russell MA, Wilson C, Taylor C, Baker CD. Effect of general practitioners' advice against smoking. Br Med J. 1979 Jul 28;2(6184):231-5. doi: 10.1136/bmj.2.6184.231. PMID 476401
- [Background] Jamrozik K, Vessey M, Fowler G, Wald N, Parker G, Van Vunakis H. Controlled trial of three different antismoking interventions in general practice. Br Med J (Clin Res Ed). 1984 May 19;288(6429):1499-503. doi: 10.1136/bmj.288.6429.1499. PMID 6426618
- [Background] Yilmaz G, Karacan C, Yoney A, Yilmaz T. Brief intervention on maternal smoking: a randomized controlled trial. Child Care Health Dev. 2006 Jan;32(1):73-9. doi: 10.1111/j.1365-2214.2006.00570.x. PMID 16398793
- [Background] Loudon K, Treweek S, Sullivan F, Donnan P, Thorpe KE, Zwarenstein M. The PRECIS-2 tool: designing trials that are fit for purpose. BMJ. 2015 May 8;350:h2147. doi: 10.1136/bmj.h2147. No abstract available. PMID 25956159
- [Background] Wu L, He Y, Jiang B, Zhang D, Tian H, Zuo F, Lam TH. Very brief physician advice and supplemental proactive telephone calls to promote smoking reduction and cessation in Chinese male smokers with no intention to quit: a randomized trial. Addiction. 2017 Nov;112(11):2032-2040. doi: 10.1111/add.13908. Epub 2017 Aug 2. PMID 28623848
- [Background] Lin PR, Zhao ZW, Cheng KK, Lam TH. The effect of physician's 30 s smoking cessation intervention for male medical outpatients: a pilot randomized controlled trial. J Public Health (Oxf). 2013 Sep;35(3):375-83. doi: 10.1093/pubmed/fdt018. Epub 2013 Mar 13. PMID 23487178
- [Background] Clinical Practice Guideline Treating Tobacco Use and Dependence 2008 Update Panel, Liaisons, and Staff. A clinical practice guideline for treating tobacco use and dependence: 2008 update. A U.S. Public Health Service report. Am J Prev Med. 2008 Aug;35(2):158-76. doi: 10.1016/j.amepre.2008.04.009. PMID 18617085
- [Background] Bobak A, Raupach T. Effect of a Short Smoking Cessation Training Session on Smoking Cessation Behavior and Its Determinants Among General Practitioner Trainees in England. Nicotine Tob Res. 2018 Nov 15;20(12):1525-1528. doi: 10.1093/ntr/ntx241. PMID 29099979
- [Background] Cheung YTD, Jiang N, Jiang CQ, Zhuang RS, Gao WH, Zhou J, Lu JH, Li H, Wang JF, Lai YS, Sun JS, Wu JC, Ye C, Li N, Zhou G, Chen JY, Ou XY, Liu LQ, Huang ZH, Ho SY, Li HCW, Su SH, Yang Y, Jiang Y, Zhu WH, Yang L, Lin P, He Y, Cheng KK, Lam TH. Physicians' very brief (30-sec) intervention for smoking cessation on 13 671 smokers in China: a pragmatic randomized controlled trial. Addiction. 2021 May;116(5):1172-1185. doi: 10.1111/add.15262. Epub 2020 Oct 5. PMID 32918512
- [Background] Wray JM, Funderburk JS, Acker JD, Wray LO, Maisto SA. A Meta-Analysis of Brief Tobacco Interventions for Use in Integrated Primary Care. Nicotine Tob Res. 2018 Nov 15;20(12):1418-1426. doi: 10.1093/ntr/ntx212. PMID 29059419
- [Background] West R, Raw M, McNeill A, Stead L, Aveyard P, Bitton J, Stapleton J, McRobbie H, Pokhrel S, Lester-George A, Borland R. Health-care interventions to promote and assist tobacco cessation: a review of efficacy, effectiveness and affordability for use in national guideline development. Addiction. 2015 Sep;110(9):1388-403. doi: 10.1111/add.12998. PMID 26031929
- [Background] Stead LF, Buitrago D, Preciado N, Sanchez G, Hartmann-Boyce J, Lancaster T. Physician advice for smoking cessation. Cochrane Database Syst Rev. 2013 May 31;2013(5):CD000165. doi: 10.1002/14651858.CD000165.pub4. PMID 23728631
- [Background] Aveyard P, Begh R, Parsons A, West R. Brief opportunistic smoking cessation interventions: a systematic review and meta-analysis to compare advice to quit and offer of assistance. Addiction. 2012 Jun;107(6):1066-73. doi: 10.1111/j.1360-0443.2011.03770.x. Epub 2012 Feb 28. PMID 22175545
- [Background] Wang L, Jin Y, Lu B, Ferketich AK. A Cross-Country Study of Smoking Cessation Assistance Utilization in 16 Low and Middle Income Countries: Data From the Global Adult Tobacco Survey (2008-2012). Nicotine Tob Res. 2016 May;18(5):1076-82. doi: 10.1093/ntr/ntv139. Epub 2015 Jun 25. PMID 26116084
- [Background] Doll R, Peto R, Boreham J, Sutherland I. Mortality in relation to smoking: 50 years' observations on male British doctors. BMJ. 2004 Jun 26;328(7455):1519. doi: 10.1136/bmj.38142.554479.AE. Epub 2004 Jun 22. PMID 15213107
- [Background] GBD 2015 Tobacco Collaborators. Smoking prevalence and attributable disease burden in 195 countries and territories, 1990-2015: a systematic analysis from the Global Burden of Disease Study 2015. Lancet. 2017 May 13;389(10082):1885-1906. doi: 10.1016/S0140-6736(17)30819-X. Epub 2017 Apr 5. PMID 28390697
- See also: Related Info — https://www.precis-2.org
- Available data/document: Study Protocol — https://www.precis-2.org/Help/Documentation/Help